CLINICAL TRIAL: NCT02342210
Title: Mindfulness Group-based Intervention for Early Psychosis: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other); London Health Sciences Centre (Other); Mindfulness Without Borders (Unknown)
Responsible Party: Principal Investigator, Arlene MacDougall, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106127
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Psychotic Disorders; Schizophrenia
Keywords: Mindfulness; Group Therapy
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-A - Immediate Intervention (Other): Immediate Mindfulness Ambassador Council for Early Psychosis (MAC-EP)
  Interventions: Behavioral: Mindfulness Ambassador Council for Early Psychosis (MAC-EP)
- Group-B - Delayed Intervention (Other): 3 month treatment as usual waitlist followed by Mindfulness Ambassador Council for Early Psychosis (MAC-EP).
  Interventions: Behavioral: Mindfulness Ambassador Council for Early Psychosis (MAC-EP)

INTERVENTIONS:
Behavioral: Mindfulness Ambassador Council for Early Psychosis (MAC-EP) — MAC is a 12-week facilitated group mindfulness intervention promoting the development of social-emotional competence in youth created by Mindfulness Without Borders (MWB; www.mwb.org). A meditative practice, mindfulness focuses one's awareness on the present, acknowledging and accepting without judging one's feelings, thoughts, or bodily sensations. Each session has a unique focus (e.g., paying attention, practicing gratitude) and consists of facilitated group learning, discussion and mindfulness skills practice. Home assignments to help reinforce specific lesson are also assigned. Although MAC has demonstrated acceptability, feasibility, and promising beneficial effects in schools, it has yet to be implemented and/or evaluated in a clinical population. Its youth-focus and emphasis on building social and emotional competencies through mindfulness, in addition to teaching core mindfulness skills make it a promising intervention for youth recovering from their first episode of psychosis.

SUMMARY:
Recent research has suggested that mindfulness-based interventions for psychosis may be effective in reducing the negative symptoms of schizophrenia (e.g., social withdrawal, lack of motivation) and the distress associated with psychotic symptoms (e.g., hearing voices) and could lead to improvements in functioning and quality of life. However these findings are based on small studies that largely consist of patients with chronic illness. Little is yet known about the use of mindfulness interventions for young people recovering from their first episode of psychosis.

The purpose of this study is to determine whether the Mindfulness Ambassador Council (MAC), a 12-week facilitated group intervention promoting mindfulness skills and the development of emotional and social competencies, is an effective, feasible, and acceptable means of treating youth in the early stages of psychotic illnesses. Although the current study is hypothesis generating in nature, based on previous investigations of Mindfulness Based Interventions for psychoses (Chadwick, 2014), we are expecting that participating in the MAC intervention will result in improvements in clinical, cognitive, functional, and health service utilization parameters. Additionally, we expect that the MAC intervention will prove to be acceptable to participants and a feasible intervention for early psychotic disorders.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the Mindfulness Ambassador Council (MAC), a 12-week facilitated group mindfulness based intervention specifically designed to promote mindfulness skills and the development of emotional and social competencies in youth, is an effective, feasible, and acceptable means of treating people in the early stages of psychotic illnesses.

We intend to randomly assign 30 patients being treated for psychotic illnesses in an early intervention program to an immediate treatment intervention or a delayed treatment intervention. Participants assigned to the immediate treatment intervention will receive the MAC intervention at the onset of the study whereas those assigned to the delay treatment intervention will receive the MAC intervention after approximately 3 months in a treatment as usual control group.

Participants will be evaluated at baseline, immediately post-intervention and at 3-month post-intervention on a number measures. MAC acceptability will be assessed through the Client Satisfaction Questionnaire and qualitative interviews, MAC feasibility will be assessed through recruitment, consent and completion rates, and MAC efficacy will be assessed with a number of clinical, social, cognitive, and mindfulness skill assessment tools as well as through changes in healthcare utilization before and after administration of the MAC intervention.

Although the current study is hypothesis generating in nature, based on previous findings of Mindfulness Based Interventions for psychoses, we are expecting that participation in the MAC intervention will result in improvements on clinical, cognitive, functional, and health service utilization parameters. Additionally, we expect that the MAC intervention will be acceptable to participants and a feasible intervention for early psychotic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants must currently be in treatment at the Prevention and Early Intervention Program for Psychosis (PEPP) for psychosis. In addition, participants must have been involved in the program for a period of less than 3 years, due to the focus of this study being on the treatment of early psychosis. Participants must be between the ages of 18 and 30 years old. Participants must be fluent in English, as determined by referring clinicians or researchers (in the case of advertisement referred participants) in order to meaningfully participate in the MAC intervention and complete the assessment tools.

Exclusion Criteria:

* Potential participants that show high levels of disorganized or disruptive behaviour (as determined by a cut off score of 4 or 5 on the Positive Formal Thought Disorder or Bizarre Behaviour items of the Scale for the Assessment of Positive Symptoms [SAPS]) such that they will not be able to meaningfully participate in the MAC intervention will be excluded from the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The Scale for Assessment of Positive Symptoms (SAPS) | Baseline, Change from Baseline in SAPS at 3 months, change from baseline in SAPS at 6 months
The Scale for Assessment of Negative Symptoms (SANS) | Baseline, Change from Baseline in SANS at 3 months, change from baseline in SANS at 6 months
The Profile of Mood States - Short Form (POMS) | Baseline, Change from Baseline in POMS at 3 months, change from baseline in POMSat 6 months
The Social Functioning Scale (SFS) | Baseline, Change from Baseline in SFS at 3 months, change from baseline in SFS at 6 months
Rosenberg Self-Esteem Scale (RSES) | Baseline, Change from Baseline in RSES at 3 months, change from baseline in RSES at 6 months
The Maryland Assessment of Recovery in People With Serious Mental Illness Scale (MARS) | Baseline, Change from Baseline in MARS at 3 months, change from baseline in MARS at 6 months
Kentucky Inventory of Mindfulness Skills (KIMS) | Baseline, Change from Baseline in KIMS at 3 months, change from baseline in KIMS at 6 months
Client Satisfaction Questionnaire - 8 Items (CSQ) | Immediately Post-Intervention
Social Interaction Anxiety Scale (SIAS) | Baseline, Change from Baseline in SIAS at 3 months, change from baseline in SIAS at 6 months
Social Perception primary subtest of the Wechsler Adult Intelligence Scale (WAIS-SP) | Baseline, Change from Baseline in WAIS-SP at 3 months, change from baseline in WAIS-SP at 6 months
Theory of Mind Task (TOMT) | Baseline, Change from Baseline in TOMT at 3 months, change from baseline in TOMT at 6 months
Stroop Colour and Word Test (STROOP) | Baseline, Change from Baseline in STROOP at 3 months, change from baseline in STROOP at 6 months
Wechsler Digit Span Subtest (WDS) | Baseline, Change from Baseline in WDS at 3 months, change from baseline in WDS at 6 months
Controlled Oral Word Association Task (COWAT) | Baseline, Change from Baseline in COWAT at 3 months, change from baseline in COWAT at 6 months
Digit Symbol Coding Task (DSCT) | Baseline, Change from Baseline in DSCT at 3 months, change from baseline in DSCT at 6 months
Hopkins Verbal Learning Task Revised (HVLT) | Baseline, Change from Baseline in HVLT at 3 months, change from baseline in HVLT at 6 months
Health Care Utilization Records Pre-Intervention | Utilization during the 6 months prior to the mindfulness intervention
Qualitative Focus-group | Immediately Post-Intervention
Health Care Utilization Records Post-Intervention | Utilization during the 6 months following the mindfulness intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arlene MacDougall, M.Sc., M.D., Principal Investigator — University of Western Ontario/London Health Sciences Centre

REFERENCES:
- [Background] Bell MD, Corbera S, Johannesen JK, Fiszdon JM, Wexler BE. Social cognitive impairments and negative symptoms in schizophrenia: are there subtypes with distinct functional correlates? Schizophr Bull. 2013 Jan;39(1):186-96. doi: 10.1093/schbul/sbr125. Epub 2011 Oct 5. PMID 21976710
- [Background] Birchwood M, Todd P, Jackson C. Early intervention in psychosis. The critical period hypothesis. Br J Psychiatry Suppl. 1998;172(33):53-9. PMID 9764127
- [Background] Buchanan RW. Persistent negative symptoms in schizophrenia: an overview. Schizophr Bull. 2007 Jul;33(4):1013-22. doi: 10.1093/schbul/sbl057. Epub 2006 Nov 10. PMID 17099070
- [Background] Chambers R, Lo BCY, Allen NB. The impact of intensive mindfulness training on attentional control, cognitive style and affect. Cognitive Therapy & Research 32: 303-322, 2008.
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Norman RM, Manchanda R, Malla AK, Windell D, Harricharan R, Northcott S. Symptom and functional outcomes for a 5 year early intervention program for psychoses. Schizophr Res. 2011 Jul;129(2-3):111-5. doi: 10.1016/j.schres.2011.04.006. Epub 2011 May 5. PMID 21549566
- [Background] Shonin E, Van Gordon W, Griffiths MD. Mindfulness-based interventions: towards mindful clinical integration. Front Psychol. 2013 Apr 18;4:194. doi: 10.3389/fpsyg.2013.00194. eCollection 2013. No abstract available. PMID 23616779
- [Background] Shonin E, Van Gordon W, Griffiths MD. Do mindfulness-based therapies have a role in the treatment of psychosis? Aust N Z J Psychiatry. 2014 Feb;48(2):124-7. doi: 10.1177/0004867413512688. Epub 2013 Nov 12. No abstract available. PMID 24220133
- [Background] Tan LB, Lo BC, Macrae CN. Brief mindfulness meditation improves mental state attribution and empathizing. PLoS One. 2014 Oct 17;9(10):e110510. doi: 10.1371/journal.pone.0110510. eCollection 2014. PMID 25329321
- [Background] Wenk-Sormaz H. Meditation can reduce habitual responding. Altern Ther Health Med. 2005 Mar-Apr;11(2):42-58. PMID 15819448
- [Background] Zeidan F, Faust M. The efffects of brief mindful training on cognitive control. In Southeastern psychological association conference, Charlotte, NC, 2008.
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- See also: Heinssen, R.K., Goldstein, A.B., & Azrin, S.T. (2014). Evidence-Based Treatments for First Episode Psychosis: Components of Coordinated Specialty Care. Recovery After An Initial Schizophrenia Episode (RA1SE). — http://www.nimh.nih.gov/health/topics/schizophrenia/raise/nimh-white-paper-csc-for-fep_147096.pdf
- See also: Mindfulness Without Borders — http://www.mwb.org